CLINICAL TRIAL: NCT05259891
Title: CAPTURE:eegCap Application in Paediatrics wiTh redUced GCS in REsus
Brief Title: eegCap Application in Paediatrics wiTh redUced GCS in REsus
Acronym: CAPTURE
Status: Completed | Type: Observational
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Dr. Deirdre Murray, Associate Professor and Consultant Paediatrician, Department of Paediatrics and Child Health and INFANT, UCC, Cork University Hospital, University College Cork
Other Study IDs: DM01/UCC21
Record Dates: First submitted 2022-02-18; First posted 2022-03-02 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Status Epilepticus; Altered Level of Consciousness; Non-epileptic Seizures; Epilepsy; Encephalopathy
Keywords: EEG; Emergency Department; Paediatrics; Reduced Glasgow Coma Scale (GCS)
MeSH Terms: conditions — Status Epilepticus; Consciousness Disorders; Seizures; Epilepsy; Brain Diseases; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Children frequently present with altered or reduced consciousness levels to emergency departments. By using EEG monitoring, subclinical seizure activity may be detected, leading to earlier pharmacological intervention and improved outcomes. Post-ictal phases that may be interpreted as seizure activity may become less over-treated. A feasibility study will ascertain if EEG monitoring can be applied successfully in this cohort, within a specified time period, obtaining minimum artefact (defined as < 25% artefact). EEG recordings will not be used to guide clinical management during this feasibility study.

DETAILED DESCRIPTION:
See study protocol attached

ELIGIBILITY:
Inclusion Criteria:

Children between 0 and 15 years and 11 months who present to Resuscitation Room, ED, CUH with a Glasgow Coma Scale (GCS) < 11 or, a reduction in baseline GCS in the case of children with significant neurodisability at baseline

Exclusion Criteria:

* Polytrauma
* Open head wounds
* Unstable airway or requirement for bag and mask ventilation, where cap application would affect clinical management

Ages: 0 Months to 176 Months | Sex: All
Age Groups: Child
Study Population: The study population is all children between 0 years and 15 years and 11 months who present to the Resuscitation room of the Emergency Department of Cork University Hospital. Children can have underlying co-morbidities ( eg neurodisability, epilepsy) or be their first time presenting to a hospital.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
The percentage of children who had EEG monitoring applied within twenty minutes and obtainment of an interpretable EEG recording with less than 25% artefact. | Anticipated 12 month study period

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre Murray, Principal Investigator — UCC and INFANT Centre
Locations (1):
- Cork University Hospital (CUH), Cork, Munster, Ireland